CLINICAL TRIAL: NCT04241640
Title: Nefopam for Post Video-Assisted Thoracoscopic Lobectomy Pain Management and the Improvement of Enhanced Recovery After Surgery (ERAS): a Randomized Controlled Trial
Brief Title: Nefopam for Post Video-Assisted Thoracoscopic Lobectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Chaowanan Khamtuikrua, Principal Investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SI 001/2020
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2023-06

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Nefopam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nefopam group[ (Experimental)
  Interventions: Drug: Nefopam 20 MG/ML
- placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nefopam 20 MG/ML — Nefopam group nefopam 20 mg during surgery and follow by 80 mg in 24 hours postoperative
  Arms: Nefopam group[
Drug: Placebo — Placebo
  Arms: placebo group

SUMMARY:
Video-assisted thoracoscopic (VATs) lobectomy is mild to moderately pain procedure. For conventional thoracotomy, there are many invasive pain control such as epidural analgesia, paravertebral block. However, for VATs, the invasive pain control somehow are too invasive. Nefopam is non-opioid painkilling medication, Serotonin, norepinephrine, dopamine reuptake inhibitor. Many study were demonstrated positive outcome of nefopam usage in many operation such as abdominal surgery, laparocopic surgery, orthopedic surgery. Nevertheless, nefopam for VATs is not well studied yet.

ELIGIBILITY:
Inclusion Criteria:

* Schedule to video-assisted thoracoscopic surgery : VATs lobectomy
* Can operate a patient-controlled analgesia (PCA) device
* No contraindication for nefopam

Exclusion Criteria:

* Epilepsy, on monoamine oxidase (MAO) inhibitors, glaucoma
* Creatinine clearance < 60 ml/min
* Liver disease: child-pugh score B or C
* Allergy to nefopam
* Chronic opioid use

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
morphine consumption in first 24 hours post-operative | 24 hours
  morphine consumption record from patient-controlled analgesia machine in 24 hours post-operative

SECONDARY OUTCOMES:
numeric pain score | 24 hours
  numeric pain score in 1, 2, 12, 24 hours after surgery
side effect of nefopam | 24 hours
  side effect of nefopam: tachycardia, sweating, nausea, vomiting, sedation

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine Siriraj hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No